CLINICAL TRIAL: NCT02986087
Title: Feto-Endoscopic Tracheal Occlusion (FETO) for Severe Congenital Diaphragmatic Hernia
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-6413
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Congenital Diaphragmatic Hernia; Pulmonary Hypoplasia; Pulmonary; Hypertension
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Fetal Tracheal Occlusion (Experimental): Fetuses with severe or moderate congenital diaphragmatic hernia will be offered fetal tracheal occlusion to increase lung growth.
  Interventions: Device: Fetal Tracheal Occlusion

INTERVENTIONS:
Device: Fetal Tracheal Occlusion — Fetuses with congenital diaphragmatic hernia with an observed to expected lung-to-head ratio of <25%, LHR <1, o/e LHR<30% (moderate), singleton pregnancy, no known other anomalies, gestational age < 29 weeks 6 days, no maternal disease, maternal age > 18 years old meet criteria to be offered tracheal occlusion. We want to test feasibility and efficacy in our center.
  Other Names: FETO; Fetal Endoluminal Tracheal Occlusion

SUMMARY:
Tracheal occlusion IDE approved by FDA for congenital diaphragmatic hernia fetuses.

DETAILED DESCRIPTION:
Fetuses with congenital diaphragmatic hernia with liver-up, and an observed to expected lung-to-head ratio of <25%, LHR <1, or a moderate category with o/e LHR <30%, singleton pregnancy, no known other anomalies, gestational age < 29 weeks 6 days (severe), gestational age < 31 weeks 6 days (moderate), no maternal disease, maternal age > 18 years old…. meet criteria to be offered fetal tracheal occlusion. We want to test feasibility and efficacy in our center.

ELIGIBILITY:
Inclusion Criteria:

* Isolated CDH with liver up
* Severe pulmonary hypoplasia with ultrasound O/E LHR <25% at the time of surgery
* Gestational age at FETO procedure 27 weeks 0 days to 29 weeks 6 days
* Moderate pulmonary hypoplasia with ultrasound O/E LHR <30% and liver-up at the time of surgery
* Gestational age at FETO procedure 30 weeks 0 days to 31 weeks 6 days in this moderate category
* Maternal age greater than or equal to 18 years
* Gestational age at enrollment prior to 29 weeks 6 days, or 31 weeks 6 days in moderate category
* Normal karyotype or FISH
* Normal fetal echocardiogram
* Singleton pregnancy
* Willing to remain in the greater Cincinnati area for remainder of pregnancy
* Family considered and decline option of termination of the pregnancy at less than 24 weeks 0 days
* Family meets psychosocial criteria

Exclusion Criteria:

* Patient < 18 years old
* Multi-fetal pregnancy
* Rubber latex allergy
* Preterm labor, cervix shortened (<15 mm) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Bilateral CDH, isolated left sided CDH with an O/E > 30%
* Additional fetal anomaly by ultrasound, MRI, or echocardiogram
* Chromosomal abnormalities
* Maternal contraindications to fetoscopic surgery or severe maternal condition in pregnancy
* Incompetent cervix with or without a cerclage
* Placental abnormalities known at time of enrollment
* Maternal HIV, Hepatits B, Hepatitis C
* Maternal uterine anomaly
* No safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change lung growth on prenatal imaging | prenatal period up to 40 weeks gestation
  Change in o/eLHR and other prenatal imaging tests

SECONDARY OUTCOMES:
Change survival in the severe congenital diaphragmatic hernia subgroup | 6 months
  Change rate of survival
Change need for ECMO therapy | 6 months
  Change need for ECMO therapy
Change pulmonary hypertension | 6 months
  Change pulmonary hypertension
Change neonatal morbidity | 1 year
  Change neonatal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Schibler, MD, Study Chair — CCHMC Oversight Data Safety Monitoring Committee
Locations (1):
- Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No